CLINICAL TRIAL: NCT05195294
Title: A Multi-center, Phase 2 Study for Autologous T Cells Transfected With mRNA Encoding HBV Antigen-specific TCR (LioCyx-M) as Monotherapy or as Combination With Lenvatinib for Advanced HBV-related Hepatocellular Carcinoma
Brief Title: Study of HBV-TCR T Cells (LioCyx-M) as Monotherapy or as Combination With Lenvatinib for HBV-related HCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lion TCR Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LTCR-HCC-3-4
Record Dates: First submitted 2021-06-03; First posted 2022-01-18 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer, Adult; Liver Cell Carcinoma
Keywords: TCR T cells; Hepatocellular Carcinoma; HBV; Hepatitis B virus
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LioCyx-M monotherapy (Experimental): Patients will receive up to 8 biweekly infusions of HBV antigen specific TCR redirected T cells (LioCyx-M).
  Interventions: Biological: LioCyx-M
- LioCyx-M + lenvatinib combinational therapy (Experimental): Patients will receive up to 8 biweekly infusions of HBV antigen specific TCR redirected T cells (LioCyx-M) with daily intake of lenvatinib.
  Interventions: Biological: LioCyx-M; Drug: Lenvatinib

INTERVENTIONS:
Biological: LioCyx-M — HBV antigen specific TCR redirected T cells
Drug: Lenvatinib — 12 mg once daily for patients ≥60 kg, 8 mg for patients <60kg by oral
  Arms: LioCyx-M + lenvatinib combinational therapy

SUMMARY:
This is an open-label and multi-center Phase 2 study to evaluate the safety and efficacy of autologous T-cells transfected with mRNA encoding Hepatitis-B virus (HBV)-antigen-specific T cell receptor (TCR) (LioCyx-M) as monotherapy or as combination with lenvatinib for the treatment of advanced HBV-related hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
2. Advanced HCC with diagnosis confirmed by histology/ cytology or clinically by AASLD criteria in cirrhotic patients.
3. Disease that is not amenable to curative surgical and/or locoregional therapies, or progressive disease after surgical and /or locoregional therapies
4. Patients who failed first-line systemic therapy for HCC
5. Serum HBsAg positivity
6. Non-cirrhotic or compensated cirrhosis Child-Pugh A (5 - 6 points)
7. HLA class 1 profile matching HLA-class I restriction element of the available T cell receptor

Exclusion Criteria:

1. Brain metastasis
2. Second primary malignancy that is clinically detectable at the time of consideration for study enrolment, except for in situ carcinoma of the cervix, non-melanoma skin carcinoma localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer and superficial bladder tumours.
3. Lack of peripheral venous or central venous access or any condition that would interfere with drug administration or collection of study samples
4. History of severe allergic anaphylactic reactions to T cell therapy products and/or lenvatinib
5. Local or loco-regional therapy of intrahepatic tumour lesions (e.g. surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) must have been completed ≥4 weeks before the first infusion of LioCyx-M.
6. Concurrent administration of any other anti-tumour therapy, including cytotoxic chemotherapy, tyrosine kinase inhibitor therapy, and immunotherapy.
7. Treatment with anticancer therapy, including investigational therapy, within 2 weeks prior to first infusion. For prior therapies with a half-life longer than 3 days, discontinuation of the therapy must have occurred at least 28 days prior to leukapheresis.
8. Treatment with other investigational therapy within 28 days prior to initiation of study treatment. Patients participating in surveys or observational studies are eligible to participate in this study.
9. Likelihood to require any immunosuppressive treatments during the period of the clinical trial (Localized steroid use should be allowed)
10. Human immunodeficiency virus (HIV) positive or active infection requiring treatment (except for HBV)
11. Significant cardiovascular disease (such as New York Heart Association (NYHA) Functional Classification Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident within 3 months prior to initiation of study treatment), unstable arrhythmia, or unstable angina
12. Uncontrolled hypertension, defined as systolic blood pressure >160 mmHg or diastolic pressure >110 mmHg, despite optimal medical management

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Assessments of adverse events/serious adverse events | Up to 4 years from study treatment initiation
  To evaluate the safety of LioCyx-M as a monotherapy and in combination with lenvatinib
Objective response rate (ORR) | Up to 4 years from study treatment initiation
  To evaluate the anti-tumor efficacy of LioCyx-M as a monotherapy and in combination with lenvatinib

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 4 years from study treatment initiation
  To evaluate the anti-tumor efficacy of LioCyx-M as a monotherapy and in combination with lenvatinib
Time to radiographic progression (TTRP) | Up to 4 years from study treatment initiation
  To evaluate the anti-tumor efficacy of LioCyx-M as a monotherapy and in combination with lenvatinib
Duration of response (DoR) | Up to 4 years from study treatment initiation
  To evaluate the anti-tumor efficacy of LioCyx-M as a monotherapy and in combination with lenvatinib
Overall survival (OS) | Up to 4 years from study treatment initiation
  To evaluate the anti-tumor efficacy of LioCyx-M as a monotherapy and in combination with lenvatinib